# Supertowel

| Improving the Supertowel: An Alternative Hand Cleaning Product fo | r |
|-------------------------------------------------------------------|---|
| Emergencies | |

Version 15/11/2019

<Amendments and previously approved versions>

SPONSOR: London School of Hygiene & Tropical Medicine

FUNDERS: The Office of U.S. Foreign Disaster Assistance (OFDA)

PRIME RECIPIENT: Real Relief

STUDY COORDINATION CENTRE: KET's Scientific Research Centre, Mumbai (India).

LSHTM ethics reference: 18006

#### PARTICIPANT INFORMATION SHEET/CONSENT FORM

# **Title of the study:** Improving the Supertowel

Principle investigators: Dr. Belen Torondel (belen.torondel@lshtm.ac.uk); Dr. Rummana Khan

Good morning/afternoon, my name is \_\_\_\_\_\_\_. I work at KET's Scientific Research Centre We are currently working on a research project with a university in England called the London School of Hygiene and Tropical Medicine (LSHTM) and an organisation called Real relief.

# What is the research project about?

In this research we will be testing a product called the Supertowel. The Super Towel has been designed as a product that can be used instead of handwashing with soap. It has been designed for humanitarian emergencies or settings where soap and water are limited.

# What is special about the Supertowel?

Even though the Supertowel may look like it is made from normal fabric, it is not. If you looked at the Magic Towel fabric under the microscope you would see an important difference. It has been treated with an 'anti-microbial shield'. This means that the material is designed to attract pathogens and when they land on the surface of the Supertowel they are caught on thousands of tiny spikes which pierce and kill the germs. There are no chemicals used to kill the germs so the Supertowel is very safe. Below you can see some images of what the Supertowel looks like under a microscope.



Above: Germs are attracted to the tiny spikes on the fabric



Above: The germs are pierced on the spikes as soon as they come into contact with them.

#### What are you being asked to do:

In this study we would like to test different hand-cleaning procedures with the Supertowel. For example we will be seeing if the Supertowel works well when it in different amounts of water, use it for different lengths of time (adding to it different amounts of water, adding to it dirty water, rubbing the hands using different times, checking if soiled Supetowel can be still effective) and compare the results obtained with washing hands with water and soap.

# Why are we inviting you to participate in the study?

We are looking for local male adult residents that are healthy and who do not have any skin conditions. We will include 16 volunteers in this study.

# Your participation is VOLUNTARY

You are free to choose whether you want to participate in this study or not. If you do agree, you are still free to withdraw participation at any time. If you decide to withdraw from the study, data associated with you will be destroyed and there will be no consequences to you or your family.

### What will happen if I decide to take part?

If you decide to take part in the study, you will be required to spend about 2-3 hours in KET's Scientific Research Centre in Mulund, Mumbai. During this time, we will get your to try hand cleaning in a variety of different ways, sometimes with the Supertowel and sometimes with bar soap. You will take part in up to 8 small handwashing tests. Each test will assess the Supertowel under different conditions. For example one test will see if it can be used with only a small amount of water, another will test whether it can be effective if used for a short period of time and others will explore whether it can be used effectively when it is visibly dirty or dipped into dirty water.

In advance of each handwashing test your hands will be artificially contaminated with a product that will not cause any harm for you (non-pathogenic E.coli). Then we will explain to you how we would like you to clean your hands. Samples will be taken before and after hand-washing in order to determine how effective the Supertowel or soap have been at removing the product that was put on your hands. Samples are taken by just pressing your fingers onto a small dish. Your participation in these experiments will be video recorded in accordance with local ethical regulations. These videos will not include your face and will not be made public and will only be viewed by the researchers involved with this study and by ethical committees if requested.

#### **Risks & Benefits**

There are no direct risks of infection to you as we will be using a contamination product for the test that cannot cause harmful effects. Upon completion of the data collection you will be provided with medicated soap in order to remove any of the product that is left on your hands. The towel has been used in previous experiments and no harmful effects have occurred.

To thank you for your time we will give you a small monetary compensation of 600 INR (to cover trip and subsistence expenses for the day you will visit the laboratory). Other than this there are no direct personal benefits of being part of this study. However, by participating in this study but you are contributing to important research that could help many others in the future.

# Privacy, anonymity and confidentiality

All the information we collect will be confidential and will be used only for the purpose of the study. We will not use your name when we share and publish the results of this study.

# **Persons to contact**

If you have any questions about the study, you can contact the Trial Manager Dr. Rummana Khan using the following contact details:

KET's Scientific Research Centre. 3rd Floor, V.G.Vaze College, Mithagar Road, Mulund (E).Mumbai -400081, India.

Mob: 9224446350

November 2019

Tel: **+91-22-21630391 Ext-213** micro@kelkarresearchcentre.org

If at any time during the study you have questions or you wish to know more about the study, you can contact the Principle Investigator on the details below:

Dr. Belen Torondel Rm 407, LSHTM Keppel Street, London WC1E 7HT

office: +442076362934

belen.torondel@lshtm.ac.uk

**Title of Project:** Improving the SuperTowel

Name of Researcher responsible for project: Dr. Belen Torondel /Dr.Rummana Khan

| Statement | | Please initial or thumbprint* each box |
|---|---|---|
| I confirm that I have read the information sheet date study. I have had the opportunity to consider the infanswered satisfactorily. <b>OR</b> | | |
| I have had the information explained to by study per<br>have had the opportunity to consider the informatio<br>answered satisfactorily. | 0 0 | |
| I understand that my participation is voluntary and without giving any reason, without my medical care | <u> </u> | |
| I understand that data collected during the study ma<br>from LSHTM and KET's Scientific Research Centre. I<br>have access to these laboratory records about my pa | give permission for these individuals to | |
| I understand that data about/from me may be share sharing directly with other researchers, and that I w information | | |
| I understand that while I participate in the laborator but that these video records will not be used unless study. | 7 - | |
| I have been given the Code of Conduct governing the a complaint should there be a breach of any of these | | |
| I agree to take part in the above named study | | |
| Printed name of participant | Signature of participant | Date |
| Printed name of impartial witness* I attest that I have explained the study information | Signature of impartial witness* accurately in to, and was u | Date nderstood to the best of |
| my knowledge by, the participant and that he/she labove named impartial witness (where applicable) | has freely given their consent to participate | |
| Printed name of person obtaining consent | Signature of person obtaining consent | Date |

[\*Only required if the participant is unable to read or write.]

# \*Code of Conduct

#### **Business and ethics**

Real Relief recognizes that the markets in which it operates are to a large extent funded by donations by governments, organizations and individuals. These donations are to mitigate the hardship caused by diseases for the individual and to improve the livelihood and outlook for households, communities and countries on levels of health, society and economy.

Bribery and other improper conduct of business profoundly impede the development of societies at every level. Real Relief recognizes that improper conduct of business may jeopardize the societal benefit intended and expressed in donations from countries, organizations and individuals, monetary and otherwise, which are fundamental to achieving the SDG 2030.

Real Relief is working with suppliers, agents, distributors and customers in

most regions of the world. We have a global perspective on matters such as human rights, working conditions, environmental matters, laws and regulations, and we comply with the same standards as would be the case if we were operating solely in Europe.

Real Relief believes that everyone has the right to a decent life – and that this vision can only be fulfilled if all stakeholders to the mission carry out their activities and obligations decently.

Real Relief seeks adherence to international standards of ethical conduct relevant to the different areas of its activities; the UN Global Compact, ILO Labor Standards, The FAO International Code.

#### **Good product**

| Quality | Real Relief will seek to ensure that its products comply with all relevant standards, |
|---|---|
| | performance and safety and that the products meet relevant specifications. |

Real Relief will conduct ongoing assessments of its products beyond the call of relevant standards to ensure they serve their purpose optimally and that all features and characteristics can be known to users and persons facilitating their use.

Safety Real Relief will seek to reduce risk to user, laborers and the environment by choice of

optimal materials, processes and formulations and seek to ensure proper labelling,

instructions and technical assistance for the correct use of its products.

Information Real Relief will seek to ensure that information accompanying or preceding its products is both sufficient and accurate and that the information is consistent with

regulatory dictate or when the information is in the form of a claim that it is based on

sound scientific evidence.

#### Sustainability

Real Relief encourage the adoption and use of environmentally sound and fully sustainable technologies, while requiring from our suppliers both voluntary approaches and a regulatory framework that nurtures innovation and economic, social and environmental accountability, all of which provide them with the necessary know-how, goods and services, equipment and organizational and managerial procedures.

#### **Good conduct**

#### Confidentially

Real Relief requires confidentiality for corporate information regarding Real Relief, its partners and affiliates. Most of the information accessed or developed in the context of business activities is proprietary. It may be company property and thus a business asset, or that of a partner in which case confidentiality shall be preserved to ensure no breach of contract and the reputation of the company. Proprietary information may never be used for personal gain during or after employment with Real Relief.

#### Corruption

Real Relief shall pursue to compete on fair grounds relating to price, product and service and shall not seek to obtain advantage in violation with local or international law.

Real Relief will not engage in any form of bribery, corruption or extortion, or otherwise seek to unjustly influence public officials or members of non-governmental organizations to obtain undue or improper advantages.

Hospitality and entertainment gifts of reasonable value are accepted as long as the above principles are observed. If any doubt in this regard a director must be consulted.

Third parties must not be used to circumvent any of these principles.

Real Relief will, when contracting agents, consultants or other third parties to act on its behalf, require full transparency and documentation in regard to contracts and fees for services, deliverables and payments, and accounting, documentation and deviations.

# **Good context**

# Environment

Real Relief shall at all times act in accordance with local regulation and law. Real Relief shall apply a precautionary approach to the environmental impact of present and future activities by assessing their potential hazard, sustainability and risk.

Real Relief shall continuously seek to improve its methods of production and product from an environmental point of view.

# Work place

Real Relief shall at all times, as a minimum, act in accordance with local regulations regarding basic wage levels, daily working hours and all other relevant regulations and laws of the individual countries where we operate.

Real Relief will not accept the use of child labour. We will specifically and continuously address this issue with all new and existing collaborators. Child labour is defined as employment of children under the age of 18 according to the main principles of the ILO's Convention concerning the minimum age of admission to employment and work.

We will demand from our collaborators that no child under the age of 18 will do any hazardous work, which is likely to jeopardize children's physical, mental or moral health or hinder their education.

Real Relief respects the freedom of association and the effective recognition of the right to collective bargaining.

#### **Good behavior**

#### Respect

(PSEA)

Real Relief observes and respects the UN Universal Declaration of Human Rights Act and will seek to promote its principles with partners within our sphere of influence. Real Relief considers any form of encouragement or assistance in the violation of these rights or knowingly ignoring such incidences as constituting a violation. Real Relief will always conduct its activities in respect of local culture and religion.

Prevention of sexual 1. Sex exploitation and abuse groun

Real Relief adheres to the core principles of the IASC Task Force on PSEA in Humanitarian Crises. The following principles therefore applies to Real Relief personnel, associates, subcontractors, suppliers or persons otherwise working under Real Relief leadership in humanitarian crises situations:

- 1. Sexual exploitation and abuse constitute acts of gross misconduct and are therefore grounds for termination of employment or contract;
- 2. Sexual activity with children (persons under the age of 18) is prohibited regardless of the age of majority or age of consent locally. Mistaken belief in the age of a child is not a defense;
- 3. Exchange of money, employment, goods, or services for sex, including sexual favors or other forms of humiliating, degrading, or exploitative behavior is prohibited. This includes exchange of assistance that is due to beneficiaries;
- 4. Sexual relationships with beneficiaries are strongly discouraged since they are based on inherently unequal power dynamics. Such relationships undermine the credibility and integrity of our work;
- 5. If anyone, working under Real Relief leadership, develops concerns or suspicions regarding sexual abuse or exploitation by a fellow worker, whether in the same organisation or not, s/he must report such concerns directly to Real Relief management 6. All staff working under Real Relief leadership are obliged to create and maintain an environment that prevents sexual exploitation and abuse and promotes the implementation of this Code of Conduct. Managers at all levels have particular responsibilities to support and develop systems that maintain this environment.

#### Conflict

Conflict of interest exists where one or both parties in a relationship receive or give unfair advantage or preferential treatment because of their interpersonal relationship.

If a Real Relief employee is unsure if the relationship with another organization or person conflicts with job performance or Real Relief's interests, the circumstances must be discussed with the relevant director.

#### Fair competition

Real Relief will adhere to local and international antitrust regulation and only participate in the market place in a fair manner and in the spirit of free competition.

#### Reporting

Obligation Real Relief encourages open discussion between management and employees regarding ethical

and compliance matters. It is the duty of every employee to report if a violation of Code of the

Ethics is believed to have occurred.

Impunity Real Relief guarantees that no person reporting a violation of its Code or international or local

law will meet in subsequent disciplinary or retaliatory action towards the reporting party.

Methods of reporting of violation may be made in person or in writing to any of the directors in

Real Relief.

# **Compliance and audit**

Company Real Relief is committed to educating its staff on the principles of its Code of Ethics as well as

training them in the compliance to the Code in their operational context.

Directors A director receiving a report of a violation must take appropriate action to remedy the offense

and its cause and register the incident and its context.

Board Real Relief's board shall annually review reports of violations of its Code and establish a

course of action to correct any systemic designs leading to faulty decision making

Improvement Real Relief will establish a system of ethical benchmarking to ensure measured

and ongoing improvement on issues related to all dimensions of its Code of Ethics and

progress towards full adherence to the provisions of the Global Compact.